CLINICAL TRIAL: NCT00423514
Title: A Phase I/II Dose Escalation Trial of Clofarabine, in Addition to Melphalan and Thiotepa as Myeloablative Regimen Followed by an Allogeneic Unmodified Hematopoietic Stem Cell Transplant From HLA-Compatible Related or Unrelated Donors for the Treatment of High Risk and/or Advanced Hematologic Malignancies
Brief Title: Clofarabine, Melphalan, and Thiotepa Followed By a Donor Stem Cell Transplant in Treating Patients With High-Risk and/or Advanced Hematologic Cancer or Other Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-125; MSKCC-06125
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2021-06

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes
Keywords: graft versus host disease; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; childhood chronic myelogenous leukemia; recurrent childhood acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; blastic phase chronic myelogenous leukemia; juvenile myelomonocytic leukemia; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; childhood acute myeloid leukemia in remission; de novo myelodysplastic syndromes; recurrent childhood acute lymphoblastic leukemia; chronic phase chronic myelogenous leukemia; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Blast Crisis; Leukemia, Myelomonocytic, Juvenile; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase | interventions — Filgrastim; Clofarabine; Melphalan; Mycophenolic Acid; Tacrolimus; Thiotepa; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- cytoreduction regimen & stem cell transplant (Experimental): This is a single arm phase I/II clinical trial to assess efficacy (the antileukemic potential and relapse rate), and safety (peri-transplant morbidity and mortality) of a novel cytoreduction regimen in preparation for allogeneic hematopoietic stem cell transplantation (HSCT).
  Interventions: Biological: filgrastim; Drug: clofarabine; Drug: melphalan; Drug: mycophenolate mofetil; Drug: tacrolimus; Drug: thiotepa; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: clofarabine
Drug: melphalan
Drug: mycophenolate mofetil
Drug: tacrolimus
Drug: thiotepa
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy, such as clofarabine, melphalan, and thiotepa, before a donor stem cell transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and mycophenolate mofetil before the transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects and best dose of clofarabine when given together with melphalan and thiotepa, followed by a donor stem cell transplant and to see how well it works in treating patients with high-risk and/or advanced hematologic cancer or other disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of clofarabine when administered with melphalan and thiotepa followed by allogeneic stem cell transplantation in patients with high-risk and/or advanced hematologic malignancies. (Phase I)
* Determine the 1-year disease-free survival of patients treated with this regimen. (Phase II)
* Determine the efficacy of this regimen, in terms of antileukemic potential and relapse rate, in these patients.

Secondary

* Evaluate the incidence and severity of nonhematologic toxicity of this regimen in these patients.
* Evaluate the incidence and severity of graft-versus-host disease in patients treated with this regimen.

OUTLINE: This is a phase I, dose-escalation study of clofarabine followed by an open-label, phase II study. Patients are stratified according to HLA-compatible donor type (related vs unrelated).

* Cytoreductive therapy: Patients receive clofarabine IV over 2 hours once daily on days -9 to -5, thiotepa IV over 4 hours on day -4, and melphalan IV over 30 minutes once daily on days -3 and -2.

Cohorts of 3-6 patients receive escalating doses of clofarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Graft-versus-host disease (GVHD) prophylaxis: Patients who undergo bone marrow or peripheral blood stem cell transplantation receive tacrolimus IV continuously over 24 hours or orally every 8-12 hours beginning on day -3 and methotrexate IV on days 1, 3, 6, and 11. Patients who undergo UCB transplantation receive tacrolimus IV continuously over 24 hours or orally every 8-12 hours beginning on day -3 and mycophenolate mofetil (MMF) IV or orally 2 or 3 times daily on days -3 to 45 followed by a taper until day 100 (unless there are signs of acute GVHD). Patients who undergo UCB transplantation without GVHD continue tacrolimus for 6 months followed by a taper and discontinued 1 year after transplantation.
* Allogeneic hematopoietic stem cell transplantation (HSCT) or allogeneic umbilical cord blood (UCB) transplantation: Patients undergo allogeneic HSCT (bone marrow or peripheral blood stem cells) or double UCB transplantation on day 0. Patients also receive filgrastim (G-CSF) IV or subcutaneously beginning on day 7 and continuing until blood counts recover.
* Maintenance therapy: Approximately 2 months after transplantation patients with ALL, M4 or M5 AML, and those transplanted with AML in bone marrow relapse receive cytarabine intrathecally (IT) monthly for up to 5 doses. Patients with a history of CNS leukemia receive cytarabine IT once monthly during months 2-12 after HSCT.

After completion of study therapy, patients are followed periodically for at least 4 years.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Acute myelogenous leukemia, meeting 1 of the following criteria:

    * In first complete remission (CR), meeting 1 of the following criteria:

      * Poor risk [no t(15,17), inv 16, or t(8,21)]
      * Not a candidate for total body irradiation (TBI)
      * Any infant in first CR
    * In second CR, meeting the following criteria:

      * All patients
    * In more than second CR OR relapsed/refractory disease, meeting the following criteria:

      * All patients
      * Blast percentage > 5% and < 25% in bone marrow (BM) at the time of stem cell transplantation (SCT)
  * Acute lymphoblastic leukemia, meeting 1 of the following criteria:

    * In first CR, meeting 1 of the following criteria:

      * Poor risk [t(9;22), t(4;11) AND no CR after 7-28 days of induction]
      * Not a candidate for TBI
      * Any infant in first CR
    * In second CR, meeting the following criteria:

      * All patients
    * In more than second CR OR relapsed/refractory disease, meeting the following criteria:

      * All patients
      * Blast percentage > 5% and < 25% in BM at the time of SCT
    * Acute undifferentiated or biphenotypic leukemia, meeting the following criteria:

      * All patients
      * Blast percentage > 5% and < 25% in BM at the time of SCT
    * Chronic myelogenous leukemia, meeting the following criteria:

      * All patients
      * In first chronic phase
    * Myelodysplastic syndrome, meeting 1 of the following criteria:

      * Primary high risk disease

        * Stage > RAEB1
      * Secondary high risk disease

        * All patients
        * Any stage
      * Juvenile myelomonocytic leukemia

        * All patients
* No doubling of peripheral blast counts within a period of 2 weeks
* No active CNS disease
* HLA-compatible donor available meeting 1 of the following criteria:

  * Related donor

    * Genotypically or phenotypically matched at ≥ 7 or 8 of HLA-A, -B, -C and -DRB1 alleles
  * Unrelated donor meeting 1 of the following criteria:

    * 8 of 8 alleles matched
    * For patients < 18 years old only: 7 or 8 alleles matched with the mismatch at only 1 HLA-A, -B, -C, or -DRB1 allele
* Two HLA-compatible unrelated cord blood (UCB) units available meeting the following criteria:

  * HLA-matched minimally at 4 of 6 HLA-A, HLA-B, and DRB1 allele

    * HLA-A and HLA-B matched at intermediate resolution by molecular technique
    * DRB1 allele matched at high resolution by molecular technique
  * Both matched UCB units with cryopreserved nucleated cell dose ≥ 1.5 x 10^7/kg

PATIENT CHARACTERISTICS:

* Karnofsky OR Lansky performance status 70-100%
* SGOT < 2 times upper limit of normal
* Bilirubin < 1.5 mg/dL (unless there is liver disease involvement)
* Creatinine normal OR creatinine clearance > 60 mL/min
* LVEF > 50% at rest OR shortening fraction ≥ 29%
* Patients with asymptomatic pulmonary disease with no prior risk factors OR symptomatic pulmonary disease with diffusion capacity > 50% of predicted (corrected for hemoglobin) are eligible
* No active uncontrolled viral, bacterial, or fungal infection
* No known HIV I or II positivity
* No known human T-cell lymphotrophic virus I or II positivity
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No hydroxyurea within the past 2 weeks
* No allogeneic or autologous stem cell transplantation within the past 6 months

Ages: 0 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2006-11-20 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farid Boulad, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Clofarabine at 20 mg/m^2/Dose x 5 + THIO-MEL; Dose Level 2: Clofarabine at 30 mg/m^2/Dose x 5 + THIO-MEL: This is a single arm phase I/II clinical trial to assess efficacy (the antileukemic potential and relapse rate), and safety (peri-transplant morbidity and mortality) of a novel cytoreduction regimen in preparation for allogeneic hematopoietic stem cell transplantation (HSCT).
Period: Overall Study
Arm/Group | Dose Level 1: Clofarabine at 20 mg/m^2/Dose x 5 + THIO-MEL | Dose Level 2: Clofarabine at 30 mg/m^2/Dose x 5 + THIO-MEL
Started | 31 | 7
Completed | 30 | 7
Not Completed | 1 | 0
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Clofarabine at 20 mg/m^2/Dose x 5 + THIO-MEL | Dose Level 2: Clofarabine at 30 mg/m^2/Dose x 5 + THIO-MEL | Total
Number analyzed (Participants) | 31 | 7 | 38
Age, Continuous [Median (Full Range); unit: years] | 17 [1 to 58] | 26 [2 to 56] | 18 [1 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 19 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 27 | 6 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 24 | 6 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: USA | 29 | 7 | 36
  United States: England | 1 | 0 | 1
  United States: Canada | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Response to Therapy
Description: * A complete response (CR) will be defined as less than 5% bone marrow blasts in the setting of a neutrophil count of >/= 1.0 K/ul and a platelet count of >/= 75,000/ul
  * A complete response except platelets (CRp) will be defined as less than 5% bone marrow blasts in the setting of a neutrophil count of >/= 1.0 K/ul and a platelet count of >/= 75,000/ul
  * A partial response (PR) will be defined as 5%-25% bone marrow blasts in the setting of a neutrophil count of >/= 1.0 K/ul and a platelet count of >/= 75,000/ul
  * A partial response except platelets (PRp) will be defined as 5%-25% bone marrow blasts in the setting of a neutrophil count of >/= 1.0 K/ul and a platelet count of >/= 75,000/ul
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Clofarabine at 20 mg/m^2/Dose x 5 + THIO-MEL | Dose Level 2: Clofarabine at 30 mg/m^2/Dose x 5 + THIO-MEL
Number analyzed (Participants) | 31 | 7
Participants
  Relapse | 1 | 0
  Complete Response | 27 | 4
  Not evaluable | 3 | 3

2. Primary Outcome: Overall Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Clofarabine at 20 mg/m^2/Dose x 5 + THIO-MEL | Dose Level 2: Clofarabine at 30 mg/m^2/Dose x 5 + THIO-MEL
Number analyzed (Participants) | 31 | 7
Participants
  Alive | 19 | 4
  Dead | 12 | 3

3. Secondary Outcome: Participants Evaluated for Early Post-transplant Regimen-related Severe Morbidity (Grade III to IV Nonhematologic Toxicity) and Mortality as Measured by the NCI Cancer Therapy Evaluation Program CTCAE v 3.0
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Clofarabine at 20 mg/m^2/Dose x 5 + THIO-MEL | Dose Level 2: Clofarabine at 30 mg/m^2/Dose x 5 + THIO-MEL
Number analyzed (Participants) | 31 | 7
Participants | 31 | 7

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dose Level 1: Clofarabine at 20 mg/m^2/Dose x 5 + THIO-MEL | Dose Level 2: Clofarabine at 30 mg/m^2/Dose x 5 + THIO-MEL
All-Cause Mortality (participants affected / at risk) | 12/31 | 3/7
Serious Adverse Events (participants affected / at risk) | 8/31 | 3/7
Other Adverse Events (participants affected / at risk) | 31/31 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Clofarabine at 20 mg/m^2/Dose x 5 + THIO-MEL (N=31) | Dose Level 2: Clofarabine at 30 mg/m^2/Dose x 5 + THIO-MEL (N=7)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0
Death not assoc w CTCAE term - Disease prog NOS (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Ileus, GI (func obstruction of bowel) (Gastrointestinal disorders) | 1 | 0
Infection, other (Infections and infestations) | 1 | 1
Liver dysfunction/failure (Hepatobiliary disorders) | 1 | 1
Metabolic/Lab - Other (specify) (Metabolism and nutrition disorders) | 1 | 0
Mucositis (Clin exam) - Oral cavity (Gastrointestinal disorders) | 1 | 1
Pneumonitis/pulm infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash; erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Secondary malig - poss related to ca txt specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Clofarabine at 20 mg/m^2/Dose x 5 + THIO-MEL (N=31) | Dose Level 2: Clofarabine at 30 mg/m^2/Dose x 5 + THIO-MEL (N=7)
ALT, SGPT (Investigations) | 20 | 5
AST, SGOT (Investigations) | 16 | 5
Alkaline phosphatase (Investigations) | 1 | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 8 | 2
Creatinine (Investigations) | 1 | 2
Fibrinogen (Investigations) | 2 | 0
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 20 | 3
Hemoglobin (Blood and lymphatic system disorders) | 30 | 7
Leukocytes (total WBC) (Investigations) | 30 | 7
Lymphopenia (Investigations) | 30 | 7
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 13 | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 30 | 7
PTT (Investigations) | 3 | 0
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 5 | 2
Platelets (Investigations) | 30 | 7
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 4 | 0
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 16 | 1
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 11 | 2
INR (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT00423514/Prot_SAP_000.pdf